CLINICAL TRIAL: NCT06598605
Title: An Intervention Program to Improve Emotion Regulation Among Parents of Children with ASD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Responsible Party: Principal Investigator, Yael Enav, Head of Emotiinal Regulation and Mentalization Lab, University of Haifa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 491/22
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-07

CONDITIONS: ASD
Keywords: ASD; mentalization; reflective function; emotional regulation
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Parental Reflective Functioning intervention Group (Experimental): Participants will attend four online psycho-educational workshop sessions via Zoom, where they will learn strategies for emotion regulation and mentalization to improve their relationship with their children on the autism spectrum.
  Interventions: Behavioral: Parental Reflective Functioning Workshop
- Waitless control group (No Intervention): Group will undergo same measurements points with no intervention.

INTERVENTIONS:
Behavioral: Parental Reflective Functioning Workshop — Four online workshop sessions via Zoom will be based on psycho-educational knowledge concerning emotional regulation and specialized in autism. The group size will be up to 15 participants, with each session lasting an hour and a half, after which participants will be asked to complete a reflective journal.
  Arms: Parental Reflective Functioning intervention Group

SUMMARY:
To examine the effectiveness of a short-term therapeutic workshop in improving reflective functioning, the belief that emotions can change, the reported use of effective emotional regulation strategies, and perceived parental self-efficacy and child behavior.

DETAILED DESCRIPTION:
The subjects will:

Answer questionnaires and clinical interviews about the relationship with their children and their mental functioning before the workshop.

The intervention group will participate in a 4-session workshop (once a week) led by an educational psychologist specializing in autism.

Answer questionnaires and clinical interviews about emotional regulation and mental functioning among their children, and about the nature of the relationship with their children after the workshop.

ELIGIBILITY:
Inclusion Criteria:

A parent aged 18 or older of a child aged 2-18 years diagnosed with ASD

Exclusion Criteria:

* A parent under the age of 18
* A parent of a child without an ASD diagnosis
* A parent of a child with ASD diagnosis under 2 years of age, or above 18 years of age

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-12-14 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Positive and negative affect scale (PANAS) | Up to 20 weeks
  The PANAS consists of 20 items, with 10 items assessing positive affect and 10 items assessing negative affect. Participants rate each item on a 5-point Likert scale ranging from 1 (very slightly or not at all) to 5 (extremely), based on how they feel over a specified time frame.

SECONDARY OUTCOMES:
Depression Assessment Questionnaire(CES-D) | Up to 20 weeks
  The CES-D consists of 20 items, each rated on a 4-point Likert scale ranging from 0 (rarely or none of the time) to 3 (most or all of the time), based on the frequency of symptoms experienced in the past week.
State-Trait Anxiety Inventory (STAI) | Up to 20 weeks
  The STAI consists of 40 items, divided into two subscales: the State Anxiety Scale (S-Anxiety) with 20 items, and the Trait Anxiety Scale (T-Anxiety) with 20 items.Each item is rated on a 4-point Likert scale. For the S-Anxiety scale, the response options range from 1 (not at all) to 4 (very much so). For the T-Anxiety scale, the response options range from 1 (almost never) to 4 (almost always).
Beck's Depression Inventory (BDI) | Up to 20 weeks
  The BDI-II consists of 21 multiple-choice items, each describing a specific symptom or attitude associated with depression. Each item is rated on a 4-point scale ranging from 0 to 3, reflecting the severity of the symptom over the past two weeks.
Interpersonal Trust Evaluation Questionnaire (ITE) | Up to 20 weeks
  The questionnaire consists of 12 items. Each item is rated on a 6-point Likert scale ranging from 1 (Strongly Disagree) to 6 (Strongly Agree).
Perceived Stress Scale (PSS) | Up to 20 weeks
  The questionnaire consists of 14 items. Respondents indicate how often they felt or thought a certain way on a scale ranging from 0 (never) to 4 (very often). Some versions may have been adapted or shortened for specific research or clinical purposes.
Mental Health Continuum-Short Form Questionnaire (MHC-SF) | Up to 20 weeks
  The Mental Health Continuum-Short Form (MHC-SF) is a psychological assessment tool used to measure positive mental health. The MHC-SF is a shorter version of the Mental Health Continuum-Long Form (MHC-LF) and is designed to assess well-being across three dimensions: emotional well-being, social well-being, and psychological well-being. Each item is rated on a 6-point Likert scale, ranging from 0 ("never") to 5 ("every day"). The responses reflect the frequency of these positive experiences over the past month. Scores are calculated for each dimension, and a total score is obtained by summing the items. Higher scores indicate higher levels of well-being.
Subjective Happiness Scale (SHS) | Up to 20 weeks
  The Subjective Happiness Scale (SHS) consists of four items that measure global subjective happiness. Respondents rate each item on a scale from 1 to 7, where 1 indicates "not at all" and 7 indicates "a great deal." The scale provides a total score, which is the sum of the four items, with higher scores indicating higher levels of subjective happiness.
Parenting Sense of Competence (PSOC) | Up to 20 weeks
  consists of a total of 17 items. These items are divided between the two subscales: Parental Satisfaction and Parental Efficacy.Each subscale consists of several items, and respondents rate each item on a 7-point Likert scale, where higher scores indicate higher levels of satisfaction or efficacy in parenting.
Parental Reflective Functioning Questionnaire (PRFQ-18) | Up to 20 weeks
  The PRFQ-18 questionnaire consists of 18 items which respondents rate each item on a 7-point Likert scale, where higher scores indicate higher levels of reflective functioning.
Emotion Regulation Questionnaire (ERQ) | Up to 20 weeks
  The ERQ consists of 10 items that assess two main strategies of emotion regulation:Cognitive Reappraisal and Expressive Suppression.Respondents rate each item on a Likert scale typically ranging from 1 (strongly disagree) to 7 (strongly agree), indicating the extent to which they engage in each strategy.
Toronto Alexithymia Scale (TAS) | Up to 20 weeks
  The TAS consisted of 20 items, though there are variations such as the TAS-20 which is commonly used. It assesses three main dimensions of alexithymia:Difficulty Identifying Feelings,Difficulty Describing Feelings, and Externally Oriented Thinking. Respondents typically rate each item on a Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree), indicating the extent to which each statement applies to them.
Parental Burnout Assessment (PBA) | Up to 20 weeks
  23-item self-report that assesses the severity of parental burnout. It consists of four subscales: emotional exhaustion (9 items); contrast with the previous parental self (5 items); feelings of being frustrated as a parent (5 items); and emotional distancing from one's children (3 items). Items are rated on a 7-point Likert scale, from 0 = never to 6 = every day.
Adaptive Behavior Assessment System, Second Edition (ABAS-II) | Up to 20 weeks
  The number of items in the ABAS-II (Second Edition) includes around 276 items across various domains and scale. The questionnaire is typically completed by a caregiver or teacher who observes the individual's behaviors over a period of time. It consists of items rated on a Likert scale or as frequency counts, depending on the specific item. Scores on the ABAS-II provide an overall picture of an individual's adaptive behavior functioning and can help in planning interventions and measuring progress.
Child Behavior Checklist (CBCL) | Up to 20 weeks
  The CBCL consists of items organized into several scales and subscales that assess behavioral and emotional problems in children. It includes two main versions:CBCL/6-18 (Child Behavior Checklist for Ages 6-18), and CBCL/1.5-5 (Child Behavior Checklist for Ages 1.5-5).
  The CBCL is typically completed by parents or caregivers who rate the frequency and intensity of various behaviors observed in the child over a specified period. Items are scored on a 3-point Likert scale (0 = Not True, 1 = Somewhat or Sometimes True, 2 = Very True or Often True).
Couples Satisfaction Index (CSI) | Up to 20 weeks
  The Couples Satisfaction Index (CSI) typically consists of 32 items that assess various dimensions of relationship satisfaction. Respondents rate on a Likert scale, typically ranging from 1 (Very Dissatisfied) to 7 (Very Satisfied). Respondents are asked to indicate their level of agreement or satisfaction with each item based on their current perceptions of their relationship.

CONTACTS AND LOCATIONS:
Overall Officials: Yael Enav, Phd, Principal Investigator — University of Haifa
Locations (1):
- University of Haifa, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Yes
All IPD excluding personal information given by participants in interview (records and transcripts), however coded information for these interview will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available beginning 2 years after publication of the primary study results and will be available for 5 years.
Access Criteria: 1. Eligibility*: Access restricted to reseachers affiliated with accredited academic institutions or healthcare organizations with relevant credentials.
  2. Application*: Sumbit application form, research roposal, and CV to the principal investigator or designated contact.
  3. Review and Approval*: Applications reviewed by the data access committee. Decision within 4-6 weeks.
  4. Conditions of Use*: Data to be used solely for the approved project. Maintain confidentiality and data security. No third-party sharing withour approval.
  5. Publicatins and Reorting*: Sumbit summary or findings within 12 months.Acknowledge original study in publications and provide copies to the principal investigator.
URL: https://drive.google.com/drive/folders/0AIp54zcFNHSBUk9PVA